CLINICAL TRIAL: NCT06868823
Title: LMWH Versus UFH as ECMO Anticoagulation in Lung Transplantation: A Prospective, Observational, and Pilot Study
Brief Title: Prospective Observational Pilot Study of LMWH Versus UFH as ECMO Anticoagulation in Lung Transplantation
Acronym: LUX-ET-LT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., Prof. M.D. Miroslav Durila, Ph.D., MHA, University Hospital, Motol
Other Study IDs: EK-704-24
Record Dates: First submitted 2025-02-21; First posted 2025-03-11 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lung Transplantation; Extracorporeal Membrane Oxygenation (ECMO); Anticoagulants and Bleeding Disorders
Keywords: Lung Transplantation; Extracorporeal Membrane Oxygenation (ECMO); Anticoagulation; Low-Molecular-Weight Heparin (LMWH); Unfractionated Heparin (UFH); Thrombosis Prevention; Bleeding Complications; Coagulation Management in Surgery; Hemorrhagic and Thrombotic Events; Perioperative Hemostasis
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UFH Anticoagulation Group: Participants in this group will receive unfractionated heparin (UFH) as the standard anticoagulation regimen during perioperative veno-arterial (V-A) ECMO support for bilateral lung transplantation.
  UFH Administration:
  A bolus of 20-40 IU/kg UFH will be administered 30 minutes before ECMO initiation.
  Continuous UFH infusion of 2-6 mL/h (dilution: 100 mg/50 mL) will be maintained.
  Coagulation Monitoring:
  ROTEM (EXTEM, INTEM, HEPTEM, FIBTEM) will be used for real-time assessment. The target CT INTEM/CT HEPTEM ratio will be maintained at 1.2-1.5 to guide anticoagulation adjustments.
  Coagulation and Hemostasis Assessments:
  Standard laboratory coagulation tests (aPTT, PT, TT, fibrinogen, FXIII, D-dimers, anti-Xa, platelet count, hemoglobin, hematocrit) will be performed at predefined timepoints.
  Point-of-care (POC) testing and thrombin generation test (TGT) will be used for additional evaluation.
- LMWH Anticoagulation Group: Participants in this group will receive low-molecular-weight heparin (LMWH) as an alternative anticoagulation strategy during perioperative veno-arterial (V-A) ECMO support for bilateral lung transplantation.
  LMWH Administration:
  A bolus of 20-40 IU/kg LMWH (Enoxaparin) will be administered 30 minutes before ECMO initiation.
  Continuous LMWH infusion of 2-6 mL/h (dilution: 100 mg/50 mL) will be maintained.
  Coagulation Monitoring:
  ROTEM (EXTEM, INTEM, HEPTEM, FIBTEM) will be used for real-time assessment. The CT INTEM/CT HEPTEM difference will be maintained at 20-30 seconds to guide anticoagulation adjustments.
  Coagulation and Hemostasis Assessments:
  Standard laboratory coagulation tests (aPTT, PT, TT, fibrinogen, FXIII, D-dimers, anti-Xa, platelet count, hemoglobin, hematocrit) will be performed at predefined timepoints.
  Point-of-care (POC) testing and thrombin generation test (TGT) will be used for additional evaluation.

SUMMARY:
The aim of this observational pilot study is to evaluate the effectiveness and safety of low-molecular-weight heparin (LMWH) compared to unfractionated heparin (UFH) as anticoagulation in perioperative ECMO during bilateral lung transplantation.

The main question this study seeks to answer is:

Does LMWH provide a safe and effective alternative to UFH for ECMO anticoagulation in lung transplantation, with reduced bleeding and thrombotic complications?

Patients undergoing bilateral lung transplantation with perioperative veno-arterial (V-A) ECMO support will be assigned to one of two anticoagulation strategies:

UFH group: Standard UFH anticoagulation monitored using ROTEM. LMWH group: Enoxaparin-based anticoagulation monitored using ROTEM. The study will assess perioperative blood loss, hemoglobin levels, transfusion needs, and thrombotic events. Additional analyses will include coagulation profile assessments using point-of-care (POC) tests, thrombin generation test (TGT), and laboratory coagulation parameters.

DETAILED DESCRIPTION:
Introduction:

Extracorporeal circulation known as "extracorporeal membrane oxygenation" (ECMO) is a method of supportive therapy for terminal respiratory failure (1-3) or temporary replacement of lung function in the perioperative period during lung transplantation (4). In the former case, it is V-V ECMO (veno-venous ECMO), while in the latter case it is V-A ECMO (veno-arterial ECMO). According to the EURO-ELSO recommendations, the use of unfractionated heparin (UFH) is recommended as anticoagulation of the ECMO set (5). However, 40-50% of patients on ECMO experience not only bleeding but also thrombotic complications (6,7). Nowadays, there is an increasing number of case reports and small studies showing that UFH is not used and instead only standard thrombosis prophylaxis with low molecular weight heparin (LMWH) is administered without signs of thrombosis in the ECMO set (8,9). ECMO has been shown to cause impaired primary hemostasis, which can be detected by devices such as the PFA 200, ROTEM-Platelet, and Multiplate. The main pathology involves platelets and to a lesser extent von Willebrand factor (vWF) (10-12). The ECMO system is a high-flow "high shear stress" system that is comparable to the arterial circulation in vivo. In this setting, the so-called "white thrombus" plays a major role in thrombosis formation. Antiplatelet drugs are commonly used to prevent thrombosis in such a system, for example in cardiology and neurology. Thus, it can be assumed that ECMO-induced impairment of primary hemostasis, specifically impaired platelet plug formation, could naturally serve as a prevention of white thrombus formation and thrombosis of the ECMO set. However, prevention of thrombosis in the venous system or on the surface of ECMO cannulae, i.e., prevention of "red thrombus formation", is still necessary because of the existence of the Virchow triad. Since the main target of action of LMWH is factor FXa and the main target of UFH is mainly factor FIIa, it can be assumed that LMWH could be sufficient to prevent thrombosis, with minimal risk of bleeding. It is important to emphasize that LMWH only minimally blocks thrombin generation and affects the conversion of fibrinogen to fibrin only to a limited extent (i.e., thrombin time - TT), unlike UFH. Moreover, ROTEM testing can be used to monitor both UFH and LMWH (13-16). A recent study published by us supports this hypothesis and suggests that the use of LMWH in patients on ECMO support may represent a safe alternative to anticoagulation or thromboprophylaxis. The study shows that its use resulted in a relatively low incidence of bleeding and thrombotic complications (17). Thus, it can be assumed that LMWH will be suitable and effective for the prevention of thrombus formation with minimal risk of bleeding, even in patients undergoing lung transplantation with perioperative ECMO support. This hypothesis is supported by studies that have found that UFH leads to higher platelet activation compared with LMWH (18-20). On the other hand, the use of activated factor FVIIa at low doses of 12 µg/kg appears to be safe (without increasing thrombotic events) and effective in reducing postoperative bleeding in cardiac surgery. Since FVIIa acts at the site of damaged endothelium, it can be assumed that relatively small doses of FVIIa will be sufficient to stop bleeding, but not so high as to cause thrombosis. In addition, it can be assumed that isolated administration of this factor may be less thrombogenic compared with other preparations that also contain factors acting on the axes of the intrinsic clotting pathway, such as prothrombin complex concentrate (PCC, contains FII, FVII, FIX, FX) or Haemate P (contains vWF and FVIII). Therefore, early administration of low-dose FVIIa may represent an effective way to minimize perioperative blood loss without increasing the risk of thrombosis (21). Another property of recombinant activated FVIIa is its ability to positively affect platelet adhesion and aggregation, which is present during ECMO support (20,22).

Aim and nature of the study:

This is a pilot observational study to prospectively compare two groups of patients with different types of anticoagulation (LMWH vs. UFH) undergoing bilateral lung transplantation with perioperative V-A ECMO support.

Hypothesis:

The use of LMWH represents a safe alternative method of ECMO anticoagulation and thromboprophylaxis that reduces the rate of bleeding and thrombotic complications compared to the current method of anticoagulation with UFH.

Methodology:

The study was approved by the Ethics Committee of Motol University Hospital. All patients enrolled in the study will sign an informed consent for participation in the study and data collection. It will be explained to the patients that there are two types of anticoagulation that are currently standardly used at Motol Hospital for patients with ECMO support. The type of anticoagulation will be determined at the discretion of the anaesthesiologist, with the aim of dividing patients as evenly as possible into different groups. Two groups of patients with different types of anticoagulation (LMWH vs. UFH) will be compared. As this is a pilot project, a total of 40 patients will be included in the study, with each group comprising 20 patients.

In case of blood loss ≥ 500 ml and ongoing bleeding, i.e. "wet operating field", the following Motol University bleeding management protocol will be initiated in both UFH and LMWH group:

* investigate PFA 200 (Col/EPI) and ROTEM (EXTEM, INTEM, FIBTEM and HEPTEM)
* in case of pathology of PFA 200 and/or CT EXTEM/CT HEPTEM - administer Novoseven at 10-30 ug/kg (recombinant activated factor VIIa)
* re-examine all ROTEM tests (EXTEM, FIBTEM, HEPTEM) and if needed normalize them:
* CT-EXTEM > 80s by administering PCC at 10-30 ug/kg
* normalise CT-HEPTEM > 240s by administering Haemate P at 10-30j/kg
* for FIBTEM pathology - administer Exacyl at 10-30 mg/kg prior to Fibrinogen administration and normalize FIBTEM MCF ≤10 mm by administering Hemocompletan at 10-30 mg/kg - or more precisely: desired MCF - current MCF x 6.25 mg/kg e.g. (10 - 4) x (6.25 x 80 kg) = 3000 mg (add 0.5 g of fibrinogen per 1 mm)
* administer platelets at EXTEM MCF ≤ 50mm and FIBTEM MCF ≥ 10mm administer 5-10 mL/kg platelets (2 TU platelets from apheresis in an adult patient) or maintain platelets ≥ 50-100 x109/L
* if bleeding continues give Factor XIII - Fibrogammin at 10-30j/kg
* if PFA Col/EPI pathology persists and bleeding continues - give Haemate P at 20-40j/kg (if not already given to correct CT INTEM)
* if bleeding continues, repeat Novoseven 10-30 ug/kg every 4 hours for a total of 3 times
* if severe bleeding continues, give full dose of Novoseven 100 ug/kg
* if bleeding does not stop - discontinue anticoagulation/thromboprophylaxis

Note:

* for blood loss over 50% of blood volume, consider Octaplas or frozen plasma (in an adult patient with blood loss over 2000-3000 ml)
* maintain normal pH, calcium, magnesium, normothermia and haematocrit ≥0.3 (required for normal primary haemostasis)
* administer 5% albumin or transfusion products as above to maintain normovolemia (try to minimise intake of other colloids or crystalloids)

Statistical analysis:

statistical program GraphPad will be used, paired t-test, p < 0.05

ELIGIBILITY:
Inclusion Criteria:

1. ⃣ Adults (≥18 years old).
2. ⃣ Patients undergoing bilateral lung transplantation with perioperative veno-arterial (V-A) ECMO support.
3. ⃣ Planned perioperative anticoagulation with either UFH or LMWH, as determined by the attending anesthesiologist.
4. ⃣ Ability to provide informed consent or consent provided by a legally authorized representative.

Exclusion Criteria:

1. ⃣ Patients receiving ECMO as a bridge to lung transplantation.
2. ⃣ Patients requiring postoperative continuation of ECMO.
3. ⃣ Patients with perioperative blood loss ≥3,000 mL.
4. ⃣ Patients undergoing lung re-transplantation.
5. ⃣ History of severe coagulopathy or bleeding disorder.
6. ⃣ Active use of antiplatelet or anticoagulant therapy (excluding study anticoagulants).
7. ⃣ Known heparin-induced thrombocytopenia (HIT).
8. ⃣ Severe liver dysfunction (Child-Pugh C) or end-stage renal disease requiring dialysis.
9. ⃣ Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients indicated for bilateral lung transplantation from the Czech Republic and Slovakia, who will undergo surgery at Motol Hospital in Prague.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative Blood Loss | Measured intraoperatively, at the end of surgery.
  Total volume of blood lost (milliliters, mL) during surgery, measured as the volume collected in suction canisters at the end of the operation, after subtracting irrigation fluids.
Change in Hemoglobin Levels during surgery and within 24 hours after surgery | Intraoperative: Change in hemoglobin from preoperative levels to the end of surgery. Postoperative: Change in hemoglobin from preoperative levels to 24 hours post-surgery.
  The difference in hemoglobin levels (g/L) measured at baseline (preoperative) and at the end of surgery and between immediate postoperative levels and after 24 hours after surgery. This outcome evaluates the extent of perioperative blood loss and its impact on oxygen-carrying capacity.
Blood Transfusion Requirements during surgery and Within 24 Hours after surgery | Intraoperative: PRBC transfusions administered during surgery. Postoperative: PRBC transfusions administered within the first 24 hours after surgery.
  The total number of packed red blood cell (PRBC) units transfused to the patient intraoperatively and within the first 24 hours postoperatively. This outcome assesses the extent of blood loss and the need for transfusion support in ECMO-supported lung transplantation.
Incidence of Thrombotic Complications during surhery and within 24 Hours postoperatively. | Intraoperative: Thrombotic events occurring during surgery. Postoperative: Thrombotic events occurring within 24 hours after surgery.
  The number of thrombotic events occurring intraoperatively and within the first 24 hours postoperatively, including ECMO circuit thrombosis, deep vein thrombosis (DVT), arterial thrombosis, pulmonary embolism (PE), myocardial infarction (MI), and ischemic stroke (CVA).
  Thrombotic complications will be identified based on clinical signs, imaging studies, and laboratory results, including:
  ECMO circuit thrombosis requiring urgent ECMO replacement. Limb ischemia due to arterial or venous thrombosis. Deep vein thrombosis (DVT) with >50% luminal obstruction, confirmed by ultrasound.
  Pulmonary embolism (PE) confirmed by CT pulmonary angiography. Myocardial infarction (MI) diagnosed based on electrocardiographic changes and cardiac biomarkers.
  Ischemic stroke (CVA) confirmed by neurological examination and brain imaging (CT/MRI).

SECONDARY OUTCOMES:
Coagulation Profile Assessed by Point-of-Care (POC) Tests | Before anticoagulation administration; 5 minutes after anticoagulation; at ≥500 mL blood loss with ongoing bleeding "wet surgical field"; 5 minutes after NovoSeven (activated FVIIa); at end of surgery before ECMO explantation; upon ICU admission
  Assessment of coagulation function using point-of-care (POC) testing, including ROTEM Sigma and PFA-200, to evaluate differences in hemostatic profiles between LMWH and UFH anticoagulation strategies during perioperative ECMO support in lung transplantation.
  ROTEM Sigma: EXTEM, INTEM, FIBTEM, HEPTEM-parameters CT (seconds), CFT (seconds), MCF (mm), ML (%) PFA-200: Col/EPI test for platelet function assessment of CT in seconds
Coagulation Profile Assessed by Thrombin Generation Test (TGT) | Before anticoagulation administration; 5 minutes after anticoagulation; at ≥500 mL blood loss with ongoing bleeding "wet surgical field"; 5 minutes after NovoSeven (activated FVIIa); at end of surgery before ECMO explantation; upon ICU admission
  Evaluation of coagulation potential and thrombin generation capacity using the Thrombin Generation Test (TGT) to compare the effects of LMWH vs. UFH on hemostatic function in ECMO-supported lung transplantation.
  Key parameters measured:
  Lag time (initiation of thrombin formation) in minutes. Peak thrombin concentration (maximum thrombin level) in nanomolar. Time to peak (speed of thrombin generation) in minutes. Endogenous thrombin potential (ETP) (total thrombin formed) in nanomolar minutes.
Coagulation Profile Assessed by Standard Laboratory Tests | Before anticoagulation administration; 5 minutes after anticoagulation; at ≥500 mL blood loss with ongoing bleeding "wet surgical field"; 5 minutes after NovoSeven (activated FVIIa); at end of surgery before ECMO explantation; upon ICU admission
  Assessment of coagulation status using standard laboratory tests to evaluate differences in hemostatic profiles between LMWH and UFH anticoagulation strategies in ECMO-supported lung transplantation.
  Blood samples will be analyzed for standard coagulation parameters, including:
  Activated partial thromboplastin time (aPTT) in seconds. Prothrombin time (PT) in seconds. Thrombin time (TT) in seconds. Fibrinogen levels in g/L. Factor XIII (FXIII) levels in %. D-dimers in mg/L FEU. Fibrin monomers (FM) in mg/L. Antithrombin activity in %. Anti-Xa level in IU/mL. Platelet count x109/L Hemoglobin in g/L.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Motol, 2nd Faculty of Medicine, Charles University in Prague and 3rd Department of Surgery, First Faculty of Medicine, Charles University, and Motol University Hospital, Lung Transplant Program, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Outcome measures (primary and secondary endpoints) Laboratory test results relevant to the study Adverse event data
Supporting Information: Study Protocol, ICF
Time Frame: from march 2025
Access Criteria: contact me to by email

REFERENCES:
- [Background] Lisman T, Adelmeijer J, Heijnen HF, de Groot PG. Recombinant factor VIIa restores aggregation of alphaIIbbeta3-deficient platelets via tissue factor-independent fibrin generation. Blood. 2004 Mar 1;103(5):1720-7. doi: 10.1182/blood-2003-07-2287. Epub 2003 Oct 30. PMID 14592825
- [Background] Brase J, Finger B, He J, Wirtz K, Stun L, McMillen R, Flynn B. Analysis of Outcomes Using Low-Dose and Early Administration of Recombinant Activated Factor VII in Cardiac Surgery. Ann Thorac Surg. 2016 Jul;102(1):35-40. doi: 10.1016/j.athoracsur.2016.01.004. Epub 2016 Feb 10. PMID 26874365
- [Background] Xiao Z, Theroux P. Platelet activation with unfractionated heparin at therapeutic concentrations and comparisons with a low-molecular-weight heparin and with a direct thrombin inhibitor. Circulation. 1998 Jan 27;97(3):251-6. doi: 10.1161/01.cir.97.3.251. PMID 9462526
- [Background] Burgess JK, Chong BH. The platelet proaggregating and potentiating effects of unfractionated heparin, low molecular weight heparin and heparinoid in intensive care patients and healthy controls. Eur J Haematol. 1997 Apr;58(4):279-85. doi: 10.1111/j.1600-0609.1997.tb01667.x. PMID 9186540
- [Background] Ajayi AA, Pharmacols FB, Cooper J, Horn EH, Rubin PC. Comparison of the effects of unfractionated heparin and the low-molecular-weight heparins dalteparin and enoxaparin on spontaneous platelet aggregation and adenosine diphosphate activity in platelets during the third trimester of pregnancy. Methods Find Exp Clin Pharmacol. 2007 Oct;29(8):539-45. doi: 10.1358/mf.2007.29.8.1116308. PMID 18040530
- [Background] Durila M, Vajter J, Garaj M, Berousek J, Lischke R, Hlavacek M, Vymazal T. Intravenous enoxaparin guided by anti-Xa in venovenous extracorporeal membrane oxygenation: A retrospective, single-center study. Artif Organs. 2025 Mar;49(3):486-496. doi: 10.1111/aor.14879. Epub 2024 Oct 3. PMID 39360891
- [Background] Yassen KA, Refaat EK, Helal SM, Metwally AA, Youssef SD, Gorlinger K. Detection and quantification of perioperative heparin-like effects by rotational thromboelastometry in living-donor liver transplant recipients: A prospective observational study. J Anaesthesiol Clin Pharmacol. 2023 Apr-Jun;39(2):285-291. doi: 10.4103/joacp.joacp_521_21. Epub 2022 Jun 15. PMID 37564856
- [Background] Rigal JC, Boissier E, Lakhal K, Riche VP, Durand-Zaleski I, Rozec B. Cost-effectiveness of point-of-care viscoelastic haemostatic assays in the management of bleeding during cardiac surgery: protocol for a prospective multicentre pragmatic study with stepped-wedge cluster randomised controlled design and 1-year follow-up (the IMOTEC study). BMJ Open. 2019 Nov 5;9(11):e029751. doi: 10.1136/bmjopen-2019-029751. PMID 31694845
- [Background] Schaden E, Schober A, Hacker S, Spiss C, Chiari A, Kozek-Langenecker S. Determination of enoxaparin with rotational thrombelastometry using the prothrombinase-induced clotting time reagent. Blood Coagul Fibrinolysis. 2010 Apr;21(3):256-61. doi: 10.1097/MBC.0b013e328337014c. PMID 20087172
- [Background] Ichikawa J, Kodaka M, Nishiyama K, Hirasaki Y, Ozaki M, Komori M. Reappearance of circulating heparin in whole blood heparin concentration-based management does not correlate with postoperative bleeding after cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):1003-7. doi: 10.1053/j.jvca.2013.10.010. Epub 2014 Feb 5. PMID 24508375
- [Background] Durila M, Vajter J, Garaj M, Smetak T, Hedvicak P, Berousek J, Vymazal T. Acquired primary hemostasis pathology detected by platelet function analyzer 200 seen during extracorporeal membrane oxygenation is sufficient to prevent circuit thrombosis: A pilot study. J Heart Lung Transplant. 2020 Sep;39(9):980-982. doi: 10.1016/j.healun.2020.05.015. Epub 2020 Jun 11. No abstract available. PMID 32591313
- [Background] Garaj M, Durila M, Vajter J, Solcova M, Marecek F, Hrachovinova I. Extracorporeal membrane oxygenation seems to induce impairment of primary hemostasis pathology as measured by a Multiplate analyzer: An observational retrospective study. Artif Organs. 2022 May;46(5):899-907. doi: 10.1111/aor.14142. Epub 2021 Dec 17. PMID 34904233
- [Background] Garaj M, Francesconi A, Durila M, Vajter J, Holubova G, Hrachovinova I. ECMO produces very rapid changes in primary hemostasis detected by PFA-200 during lung transplantation: An observational study. J Heart Lung Transplant. 2024 Nov;43(11):1771-1776. doi: 10.1016/j.healun.2024.07.012. Epub 2024 Jul 20. PMID 39038564
- [Background] Gratz J, Pausch A, Schaden E, Baierl A, Jaksch P, Erhart F, Hoetzenecker K, Wiegele M. Low molecular weight heparin versus unfractioned heparin for anticoagulation during perioperative extracorporeal membrane oxygenation: A single center experience in 102 lung transplant patients. Artif Organs. 2020 Jun;44(6):638-646. doi: 10.1111/aor.13642. Epub 2020 Feb 18. PMID 31951030
- [Background] Lee YY, Baik HJ, Lee H, Kim CH, Chung RK, Han JI, Joo H, Woo JH. Heparin-free veno-venous extracorporeal membrane oxygenation in a multiple trauma patient: A case report. Medicine (Baltimore). 2020 Jan;99(5):e19070. doi: 10.1097/MD.0000000000019070. PMID 32000456
- [Background] Chung M, Cabezas FR, Nunez JI, Kennedy KF, Rick K, Rycus P, Mehra MR, Garan AR, Kociol RD, Grandin EW. Hemocompatibility-Related Adverse Events and Survival on Venoarterial Extracorporeal Life Support: An ELSO Registry Analysis. JACC Heart Fail. 2020 Nov;8(11):892-902. doi: 10.1016/j.jchf.2020.09.004. PMID 33121701
- [Background] Nunez JI, Gosling AF, O'Gara B, Kennedy KF, Rycus P, Abrams D, Brodie D, Shaefi S, Garan AR, Grandin EW. Bleeding and thrombotic events in adults supported with venovenous extracorporeal membrane oxygenation: an ELSO registry analysis. Intensive Care Med. 2022 Feb;48(2):213-224. doi: 10.1007/s00134-021-06593-x. Epub 2021 Dec 18. PMID 34921625
- [Background] McMichael ABV, Ryerson LM, Ratano D, Fan E, Faraoni D, Annich GM. 2021 ELSO Adult and Pediatric Anticoagulation Guidelines. ASAIO J. 2022 Mar 1;68(3):303-310. doi: 10.1097/MAT.0000000000001652. PMID 35080509
- [Background] Martin AK, Mercier O, Fritz AV, Gelzinis TA, Hoetzenecker K, Lindstedt S, Marczin N, Wilkey BJ, Schecter M, Lyster H, Sanchez M, Walsh J, Morrissey O, Levvey B, Landry C, Saatee S, Kotecha S, Behr J, Kukreja J, Dellgren G, Fessler J, Bottiger B, Wille K, Dave K, Nasir BS, Gomez-De-Antonio D, Cypel M, Reed AK. ISHLT Consensus Statement on the Perioperative use of ECLS in Lung Transplantation: Part II: Intraoperative Considerations. J Heart Lung Transplant. 2026 Jan;45(1):e35-e62. doi: 10.1016/j.healun.2024.08.027. Epub 2024 Oct 23. PMID 39453286
- [Background] Zhou AL, Jennings MR, Akbar AF, Ruck JM, Oak A, Kalra A, Larson EL, Casillan AJ, Ha JS, Merlo CA, Bush EL. Utilization and outcomes of nonintubated extracorporeal membrane oxygenation as a bridge to lung transplant. J Heart Lung Transplant. 2025 Apr;44(4):661-669. doi: 10.1016/j.healun.2024.10.021. Epub 2024 Oct 30. PMID 39486773
- [Background] Dhanani Z, Gupta R. The Management of Interstitial Lung Disease in the ICU: A Comprehensive Review. J Clin Med. 2024 Nov 6;13(22):6657. doi: 10.3390/jcm13226657. PMID 39597801
- [Background] Basta MN. Severe Acute Respiratory Distress Syndrome in an Adult Patient With Human Metapneumovirus Infection Successfully Managed With Veno-Venous Extracorporeal Membrane Oxygenation. Semin Cardiothorac Vasc Anesth. 2025 Mar;29(1):74-81. doi: 10.1177/10892532241301195. Epub 2024 Nov 19. PMID 39561244